CLINICAL TRIAL: NCT00200135
Title: Financial and Clinical Impact of Repeal of the Pennsylvania Helmet Law: A Multi-Center Prospective Study Comparing Helmeted and Non-Helmeted Motorcycle Accident Victims
Brief Title: Financial and Clinical Impact of Repeal of the Pennsylvania Motorcycle Helmet Law
Status: Completed | Type: Observational
Sponsor: Memorial Medical Center (Other)
Responsible Party: Stephen L Miller, MD,FACS/ Director, Trauma Services, Memorial Medical Center
Other Study IDs: MMC 04-18
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Craniocerebral Trauma; Facial Injuries
Keywords: motorcycle accident; helmet; traumatic brain injury; financial burden
MeSH Terms: conditions — Craniocerebral Trauma; Facial Injuries; Brain Injuries, Traumatic; Financial Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Treated and released from ED (minor injuries)
- 2: Trauma, admitted to the hospital (injured)
- 3: Fatalities reported by the coroner (deaths)
- 4: Reported by the police (No medical treatment)

SUMMARY:
The purpose of this study is to find out how many helmeted versus non-helmeted motorcycle accident victims (MCA) sustain head and/or face injuries. Also, we will find out how much it costs to get medical care for head and face injuries in helmeted versus non-helmeted motorcycle victims. Finally, we will compare how long it takes helmeted versus non-helmeted motorcycle victims with face and head injuries to return to work.

DETAILED DESCRIPTION:
This is a prospective, quasi-experimental research study that will compare clinical outcomes of helmeted versus non-helmeted motorcycle victims admitted to trauma centers, as well as victims treated and released from emergency departments.

The primary objective of this study is:

* To determine if the financial charges and ratio of cost to charges (RCC), including acute hospitalization, rehabilitation or skilled care, outpatient care, and time to return to work (implying lost wages) is different between helmeted versus non-helmeted motorcyclists with head or face injuries

Secondary objectives include:

* To determine if inpatient mean total acute care and downstream charges and RCC are higher for non-helmeted versus helmeted motorcycle victims admitted to three Pennsylvania trauma centers with head and face injuries
* To determine the mean time of return to full duty work (at previous level of employment) is shorter for helmeted or non-helmeted motorcycle victims admitted to three Pennsylvania trauma centers with head and face injuries
* To determine if non-helmeted or helmeted motorcycle victims admitted to three Pennsylvania trauma centers have increased incidence and severity of head and face injuries
* To determine the incidence and severity of non-helmeted motorcycle accident victims is higher than helmeted counterparts treated and released from emergency departments for face and head injuries
* To determine if non-helmeted motorcycle victims die at scene or in emergency departments (from head and face injuries) more often than helmeted motorcycle victims
* To determine if more helmeted or non-helmeted motorcycle accident victims require no immediate medical care for head and face injuries

ELIGIBILITY:
Inclusion Criteria:

* All English speaking drivers/passengers of motorcycle accidents, 18 years or older, with head or face injuries served by participating study trauma centers, emergency departments or coroners.
* All English speaking drivers/passengers of motorcycle accidents, 18 years of age or older, served by Pennsylvania police but did not require acute medical services.

Exclusion Criteria:

* Non-English speaking
* Served by trauma center, emergency department or coroner, but without haed or face injury
* Less than 18 years of age
* Moped accidents
* Motorized bicycle accidents
* Parked motorcycle accidents
* Off road motorcycle accidents, not on a public street or highway
* Dirtbike or motorcross accidents, involving vehicles not licensed for highway use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 helmeted and 60 unhelmeted motorcycle riders in each cohort
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Miller, MD, FACS, Principal Investigator — Memorial Medical Center
Locations (2):
- United States (2):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Memorial Medical Center, Johnstown, Pennsylvania